CLINICAL TRIAL: NCT01820975
Title: The Manipulation of Dietary Protein Intake on the Anabolic Response in Healthy Young Men
Brief Title: Manipulation of Dietary Protein and the Anabolic Response
Acronym: PRO-ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 12-3-067
Record Dates: First submitted 2013-03-18; First posted 2013-03-29 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2015-05

CONDITIONS: Focus: Anabolic Response to Food Intake in Young Individuals; Condition Relevance: Skeletal Muscle Health, Sarcopenia
Keywords: Muscle protein synthesis; Dietary protein
MeSH Terms: conditions — Sarcopenia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High protein intake (Experimental): High protein intake: large bolus of protein in teh diet the day before testing
  Interventions: Dietary Supplement: High protein intake
- No protein intake (Placebo Comparator): No protein in the diet the day before testing
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Dietary Supplement: High protein intake
  Arms: High protein intake
Other: Placebo comparator — No protein intake
  Other Names: control group
  Arms: No protein intake

SUMMARY:
In the present study, the effect of habitual dietary protein on the anabolic response will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged between 18-35 years
* Healthy, recreationally active
* BMI < 30 kg/m2

Exclusion Criteria:

* Smoking
* Allergies to milk proteins (whey or casein)
* Vegetarians
* Diagnosed GI tract diseases
* Female
* Arthritic conditions
* A history of neuromuscular problems
* Previous participation in amino acid tracer studies
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein fractional synthetic rate following protein ingestion | 3 hours
  The ability of the muscle to synthesise new proteins will be assessed over a 3 h period following protein ingestion and will be compared between groups. This only occurs on one occasion.

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356